CLINICAL TRIAL: NCT07227051
Title: Optimizing Self-Monitoring Feedback Delivery for the Treatment of Overweight and Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Virginia (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00135066; R01DK140099 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; Obesity (Disorder)
Keywords: weight loss; self-monitoring; smartphone app; lifestyle intervention; digital health; mHealth; physical activity; dietary change; e-scale; wearables; activity monitor
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Micro-randomized Factorial. Under a 2x2x2x2 factorial design, participants will be randomized each week for 16 weeks to one of 16 conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self Monitoring Feedback (Experimental): Participants enrolled in the Feedback Optimization trial will be asked to complete a 60-minute Weight Loss 101 session and to track their dietary intake, physical activity, and weight each day using study-provided tools. After the first week of self-monitoring (used as a run-in), participants will be provided with weekly feedback messages. The focus and content of these messages will vary, based on a 2x2x2x2 factorial design.
  Interventions: Behavioral: Feedback on Calorie Goal Attainment; Behavioral: Feedback on Dietary Quality; Behavioral: Feedback on Physical Activity Goal Attainment; Behavioral: Goal Setting Prompt

INTERVENTIONS:
Behavioral: Feedback on Calorie Goal Attainment — Feedback composed by a study interventionist that focuses on the participant's progress toward meeting their caloric intake goal.
Behavioral: Feedback on Dietary Quality — Feedback composed by a study interventionist that provides comments on specific dietary choices that may impact weight loss success.
Behavioral: Feedback on Physical Activity Goal Attainment — Feedback composed by a study interventionist that focuses on the participant's progress toward meeting their physical activity goal.
Behavioral: Goal Setting Prompt — An open-text goal setting prompt, composed by the study interventionist, that encourages the participant to set a behavioral goal for the following week.

SUMMARY:
The purpose of this research study is to learn how to best provide weekly feedback on individual progress toward intervention goals during a weight loss program.

DETAILED DESCRIPTION:
The goal of this micro-randomized factorial trial is to learn how to best deliver self-monitoring feedback during a behavioral weight management intervention. All study participants will be provided with a "Weight Loss 101" session that provides weight loss education and behavioral skills training. At this meeting, participants will be taught how to use study-provided tools to self-monitor their dietary intake, physical activity, and weight. At the end of each week of the intervention, participants will receive an interventionist-composed feedback message based on their self-monitoring data. Every message will contain feedback about how often the participant self-monitored their dietary intake, physical activity, and weight (that is, the number of days each week that the participant monitored each) along with a message about their weight trajectory. Participants will be randomized each week to receive (or not receive) four additional feedback components each week.

The main questions that this study aims to answer are:

* which of the four additional feedback components improve adherence to self-monitoring, intervention goals, and weight loss the week after they are received?
* are there any differences in message impact depending on the person receiving the message (for example, do some messages work better for younger versus older participants) or their context (for example, are certain messages more or less helpful depending on how well the person is doing in the program)?

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* BMI greater than or equal to 25.0 kg/m2
* Weight less than or equal to 175 kg (due to scale limit)
* Own a smartphone compatible with Fitbit (e.g., an Apple iPhone running iOS 16.4 or higher or Android smartphone running Android 11 or higher) with a cellular and data plan

Exclusion Criteria:

* Weight greater than 175 kg (due to a weight limit of the study-provided scale)
* Smartphone device owned deemed incompatible with the Fitbit App
* History of bariatric surgery or plans to obtain bariatric surgery during the study period
* Current use of weight loss medications, or use of weight loss medications in the 6 months prior to initial pre-screening
* Currently participating in a weight-loss program
* Weight loss of greater than or equal to 10 lbs in the 6 months prior to initial pre-screening
* Physical limitations that prevent walking at a brisk pace for at least 10 minutes without stopping
* Use of a pacemaker or other implanted medical device
* Currently pregnant
* Currently breastfeeding
* Less than 1-year post-partum
* Plans to become pregnant within the study period
* Lack of written confirmation that the potential participant has discussed study participation with their physician if they have been diagnosed with diabetes, hypertension, or has have a history of coronary heart disease
* One or more study participants living in the household (enrollment limited to one participant per household)
* Medical conditions that contraindicate weight loss or prevent completion of the study (e.g., current diagnosis of cancer or terminal illness, dementia, etc.)
* Recent (in the past 6 months) changes in medications that affect weight
* Self-reported eating disorder within past 5 years
* Unable to complete the 17-week study (due to plans to relocate during the study period, etc.)
* Unable or unwilling to provide informed consent
* Unable to read English at the 5th grade level
* Unwilling to accept random assignment
* Unable or unwilling to download the study smartphone application, wear the physical activity monitor, or use the study e-scale
* Failure to complete baseline assessment measures
* Failure to complete at least 4 out of 6 days of self-monitoring dietary and weight self-monitoring during the behavioral run-in period
* Any other condition(s) which, in the opinion of the Principal Investigator, would adversely affect participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Weight change | 7 days
  Fitted model values will then be used to estimate the slope of weight change from day 1 (the day a feedback message is received) to day 7 of each week, with positive values representing weight gain and negative values representing weight loss.

SECONDARY OUTCOMES:
Frequency of self-monitoring weight | 7 days
  Frequency of self-monitoring weight will be defined as the number of days (0-7) for the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7) that a participant has a valid (non-outlier) e-scale weight.
Frequency of self-monitoring dietary intake | 7 days
  A valid "day" of self-monitoring dietary intake will be defined as ≥ 800 kcal, consistent with prior research. Frequency of self-monitoring dietary intake will be defined as the number of valid days (0-7) recorded the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7).
Total caloric intake | 7 days
  Total caloric intake will be calculated by summing calories consumed the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7).
Calorie goal attainment | 7 days
  Calorie goal attainment for each day during the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7) will be calculated as [TOTAL KCAL INTAKE FOR THE DAY] - [CALORIE GOAL]. Difference scores for the 7 days will be averaged over the week to assess overall adherence to the caloric intake goal during that study week.
Frequency of self-monitoring physical activity | 7 days
  Frequency of self-monitoring physical activity will be defined as the number of "valid" days (0-7) of Fitbit use the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7).
Physical activity minutes | 7 days
  Total minutes of physical activity will be calculated by summing each days' total "active zone minutes" during the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7)
Physical activity goal attainment | 7 days
  Physical activity goal attainment for each day of the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7) will be calculated as [TOTAL PHYSICAL ACTIVITY MINUTES] - [PHYSICAL ACTIVITY GOAL]. Difference scores for the 7 days will be averaged over the week to assess overall adherence to the physical activity goal during that study week

OTHER OUTCOMES:
Time to compose intervention messages (intervention costs) | through study completion, an average of 7 days
  Interventionists will log the time needed to compose each message (including a starting time and an ending time for each message) in our administrative dashboard

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Ross, Ph.D., M.P.H., Principal Investigator — Aurora Research Institute LLC; Rebecca A. Krukowski, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- Advocate Aurora Research Institute, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual-level participant data will be de-identified and made available: (1) within one year from the final outcome assessment date, (2) at the time of publication of peer-reviewed manuscript(s) based on these data, or (3) at the end of the award, whichever is soonest. Study data will be shared via the Zenodo data repository at https://zenodo.org/. Analytic code will be made publicly available via Supplementary files for any publications and/or via Zenodo through a Zenodo-GitHub link. Study protocol, informed consent form, statistical analysis plan will also be available to be shared via clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified, individual-level participant data will be made available: (1) within one year from the final outcome assessment date, (2) at the time of publication of peer-reviewed manuscript(s) based on these data, or (3) at the end of the award, whichever is soonest.
Access Criteria: Data will be made available via the Zenodo data repository (https://zenodo.org).
URL: https://zenodo.org